CLINICAL TRIAL: NCT03444051
Title: Comparison of the 20-gauge Procore® and 22-gauge Acquire® Needles for Endoscopic Ultrasound-guided Fine Needle Biopsy (EUS-FNB) of Solid Pancreatic or Peripancreatic Masses: an Observational Study.
Brief Title: Comparison of Two Endoscopic Biopsic Needles for Pancreatic Tumors
Acronym: Mousquetaires
Status: Completed | Type: Observational
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, KARSENTI, principal investigator, Société Française d'Endoscopie Digestive
Other Study IDs: Mousquetaires
Record Dates: First submitted 2018-02-18; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Pancreatic Tumor; Puncture
Keywords: EUS-FNB; comparative study
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 20-gauge Procore®: Between March and December 2017, 68 EUS-FNB were consecutively performed in our unit for a pancreatic or peripancreatic mass. The choice of the needle depended upon the availability at the time of admission:
  34 punctures were performed with a 20-gauge Procore® during the period study
  Interventions: Procedure: EUS-FNB with 20-gauge Procore® needle
- 22-gauge Acquire®: Between March and December 2017, 68 EUS-FNB were consecutively performed in our unit for a pancreatic or peripancreatic mass. The choice of the needle depended upon the availability at the time of admission:
  34 punctures were performed with a 22-gauge Acquire® during the period study
  Interventions: Procedure: EUS-FNB with 22-gauge Acquire® needle

INTERVENTIONS:
Procedure: EUS-FNB with 20-gauge Procore® needle — Puncture of a pancreatic or peripancreatic mass under Endoscopic Ultrasonography, with a 20-gauge Procore® needle
  Groups: 20-gauge Procore®
Procedure: EUS-FNB with 22-gauge Acquire® needle — Puncture of a pancreatic or peripancreatic mass under Endoscopic Ultrasonography, with a 22-gauge Acquire®
  Groups: 22-gauge Acquire®

SUMMARY:
This observational study compared quality of histological sampling of pancreatic EUS-FNB with the 20-gauge Procore® and 22-gauge Acquire® needles. In total, 68 patients were recruited. Histological diagnosis was achieved and a histological core biopsy was obtained in 82% of patients (28/34) in the 20-gauge Procore® group and 97% of patients (33/34) in the 22-gauge Acquire® group (P=0.1). Core biopsy specimens obtained were significantly longer with the 22-gauge Acquire® needle with a mean cumulative length of tissue core biopsies per needle pass of 4,33±3,46mm vs. 7,9±4,35mm for the 20-gauge Procore® (P<0,01). Reproducibility of this simple histological criterion was validated in intra and inter-observer.

DETAILED DESCRIPTION:
Between March and December 2017, 68 EUS-FNB were consecutively performed in our unit for a pancreatic or peripancreatic mass. The choice of the needle depended upon the availability at the time of admission: 34 punctures were performed with a 20-gauge Procore®, and 34 with a 22-gauge Acquire®. Histological material was studied in a blinded manner with respect to the needle, and cumulative length of tissue core biopsies per needle pass was determined. Intra and inter-observer variability of this criterion was then evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients ≥18 who were referred for EUS-FNB for solid pancreatic or peripancreatic mass were included

Exclusion Criteria:

* non-accessible pancreatic mass because of history of Billroth II or Roux-en-Y reconstruction
* coagulation disorders (such as partial thromboplastin time >42 seconds, prothrombin time [Quick value] <50%, platelet count <50 000/mm³), treatment with clopidogrel, pregnancy.
* patients <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients ≥18 who were referred for EUS-FNB for solid pancreatic or peripancreatic mass were included. The use of EUS-FNB needle was determined during EUS if the examination confirmed the presence of a pancreatic or peri-pancreatic non-hyper-vascular mass (on Doppler examination).
  According to the period of admission, the 20-gauge Procore® (Wilson Cook Medical, Winston-Salem, NC) and 22-gauge Acquire® needles (Boston Scientific Natick, MA) were alternatively available depending on the order (made in batches of 5 units). So, patients were included either in the 20-gauge Procore® group or the 22-gauge Acquire® group.
  Patients could be switched via a crossover procedure to a second EUS-FNB with the competitive needle if the first one failed to give histologic mass characterization: failure was recorded to the first needle group, and the second EUS-FNB performed with the alternate needle was recorded in the other group.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
pancreatic mass anatomopathological characterization | in the 7 days after procedure
  pancreatic mass anatomopathological characterization, presence of histological sampling and cumulative length of tissue core biopsies per needle pass.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique PARIS-BERCY, Charenton-le-Pont, France

IPD SHARING:
Plan to Share IPD: No